CLINICAL TRIAL: NCT00853307
Title: A Phase 2 Study of MLN8237, a Novel Aurora A Kinase Inhibitor, in the Treatment of Patients With Platinum-Refractory or Platinum-Resistant Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Carcinoma
Brief Title: MLN8237 for Treatment of Participants With Ovarian, Fallopian Tube, or Peritoneal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C14006; 2008-006979-72 (EudraCT Number); U1111-1187-6616 (Registry Identifier: WHO)
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Ovarian Carcinoma
Keywords: Drug therapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alisertib 50 mg (Experimental): Alisertib 50 mg, capsules, orally, twice daily for 7 days, followed by 14-day washout period in 21-day cycles until disease progression or unacceptable treatment-related toxicity (Up to 26 Cycles).
  Interventions: Drug: Alisertib

INTERVENTIONS:
Drug: Alisertib — Alisertib capsules
  Other Names: MLN8237

SUMMARY:
The purpose of this study is to evaluate the anti-tumour activity of alisertib (MLN8237) in the treatment of participants with platinum-refractory or platinum-resistant epithelial ovarian, fallopian tube, or primary peritoneal carcinomas.

DETAILED DESCRIPTION:
The drug being tested in this study is called alisertib (MLN8237). Alisertib is being tested to treat people who have platinum-refractory or platinum-resistant epithelial ovarian, fallopian tube, or primary peritoneal carcinoma. This study looked at the antitumor activity by response rate who would take alisertib.

The study enrolled 31 patients. Participants were categorized as per the disease state into 2 categories, refractory and resistant. Participants received:

• Alisertib 50 mg

All participants took alisertib 50 mg capsules every 12 hours each day for 7 days followed by a 14-day rest period in a 21-day cycle (up to 26 cycles).

This multi-center trial was conducted in France, Poland and the United States. The overall time to participate in this study was 12 months, unless it is determined that a participant would benefit from continued therapy beyond 12 months. Participants made multiple visits to the clinic, and were contacted up to a maximum of every 12 weeks up to 12 months after last dose of study drug for follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants 18 years or older.
2. Histologically or cytologically confirmed epithelial ovarian, fallopian tube, or primary peritoneal carcinoma.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
4. Postmenopausal at least 1 year, OR

   * Surgically sterile, OR
   * If childbearing potential, agree to 2 effective methods of nonhormonal contraception, or agree to completely abstain from heterosexual intercourse.
5. Able to provide written informed consent.
6. Within 7 days before study:

   * Absolute neutrophils (ANC) ≥ 1,500/μL
   * Platelets ≥100,000/ μL
   * Total bilirubin must be < 1.5 times upper limit of the normal (ULN)
   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) must be ≤ 2.5 times the ULN. AST and ALT may be elevated up to 5 times the ULN if ascribed to metastatic liver disease.
   * Creatinine clearance ≥ 30 mL/minute
7. Platinum-refractory or -resistant disease.
8. Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) OR Cancer antigen (CA) 125 level of > 40 units/mL AND clinical evidence disease.
9. Recovered from effects of prior therapy.

Exclusion Criteria:

1. Pregnant or lactating.
2. Serious illness that could interfere with protocol completion.
3. Investigational treatment 28 days prior to first dose.
4. Maximum 4 prior systemic therapies: 2 platinum-based, 1 nonplatinum cytotoxic, 1 biological.
5. Known Central Nervous System metastases.
6. Prior allogeneic bone marrow or organ transplantation.
7. Radiotherapy within 21 days prior to first dose.
8. Radiotherapy to > 25% bone marrow.
9. Major surgery or infection requiring systemic antibiotic therapy within 14 days prior to first dose.
10. Inability to swallow orally administered medication.
11. Diagnosis or treatment of another malignancy within 2 years preceding first dose of study drug except nonmelanoma skin cancer or in situ malignancy completely resected.
12. Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-03-23 (Actual); Primary Completion 2009-11-23 (Actual); Study Completion 2011-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Summit Medical Group, Berkeley Heights, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 17 investigative sites in France, Poland and the United States from 23 March 2009 to 27 January 2011.
Pre-assignment Details: Participants with a diagnosis of Platinum-refractory and Platinum-resistant epithelial ovarian, fallopian tube, or primary peritoneal carcinoma received 50 mg alisertib twice daily for 7 days in 21-day cycles.
Groups:
- Alisertib 50 mg (Platinum-Refractory): Alisertib 50 mg, capsules, orally, twice daily for 7 days, followed by 14-day washout period in 21-day cycles until disease progression or unacceptable treatment-related toxicity (Up to 26 Cycles). Platinum-refractory disease is characterized by a lack of response, progression, or recurrence of disease during a course of platinum-based therapy.
- Alisertib 50 mg (Platinum-Resistant): Alisertib 50 mg, capsules, orally, twice daily for 7 days, followed by 14-day washout period in 21-day cycles until disease progression or unacceptable treatment-related toxicity (Up to 26 Cycles). Platinum-resistant disease is characterized by progression or recurrence of malignant disease within 6 months after completion of a platinum-based regimen.
Period: Overall Study
Arm/Group | Alisertib 50 mg (Platinum-Refractory) | Alisertib 50 mg (Platinum-Resistant)
Started | 6 | 25
Completed | 4 (Completed = participants who completed the study treatment.) | 20
Not Completed | 2 | 5
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Reason Not Specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population is defined as all participants who receive any amount of alisertib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alisertib 50 mg (Platinum-Refractory) | Alisertib 50 mg (Platinum-Resistant) | Total
Number analyzed (Participants) | 6 | 25 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (15.38) | 56.6 (14.19) | 57.0 (14.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 25 | 31
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 6 | 24 | 30
  Asian | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 3 | 22 | 25
  Not Reported | 2 | 2 | 4
Primary diagnosis [Number; unit: participants]
  Epithelial Ovarian | 5 | 20 | 25
  Fallopian Tube | 0 | 1 | 1
  Primary Peritoneal Carcinoma | 1 | 4 | 5
Years Since Initial Diagnosis [Mean (Standard Deviation); unit: years] | 1.59 (0.736) | 2.26 (1.448) | 2.13 (1.356)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — ECOG performance is defined as: 0=Normal activity (fully active, able to carry on all predisease performance without restriction); 1=Symptoms but ambulatory (restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature); 2=In bed <50% of the time (ambulatory and capable of all self-care, but unable to carry out any work activities); 3=In bed >50% of the time (capable of only limited self-care); 4=100% bedridden (completely disabled, cannot carry on any selfcare, totally confined to bed or chair).
  participants
    ECOG Performance Status = 0 | 2 | 18 | 20
    ECOG Performance Status = 1 | 4 | 7 | 11
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 162.0 (4.83) | 160.9 (7.76) | 161.0 (7.34)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 65.16 (9.638) | 68.22 (17.227) | 67.63 (15.951)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: meter (m)^2] — Body Surface Area = square root [height (cm)*weight (kg) / 3600 ].
  meter (m)^2 | 1.72 (0.167) | 1.72 (0.223) | 1.72 (0.212)

OUTCOME MEASURES:

1. Primary Outcome: Combined Best Overall Response Rate Based on Investigator Assessment
Description: Combined objective response rate is defined as the percentage of participants with Complete Response (CR) + Partial Response (PR) as assessed by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1 or response by Cancer antigen (CA) 125 criteria. According to RECIST: CR is defined as disappearance of all target lesions and PR is defined as 30% decrease in the sum of the longest diameter of target lesions. CA 125 response criteria is defined as either: A 50% decrease from 2 initially elevated samples; the sample demonstrating the 50% decrease must have been confirmed by a fourth sample 28 days later (a total of 4 samples required) or A serial decrease of > 75% over 3 samples; the third sample was to be obtained 28 days after the second (a total of 3 samples required).
Time Frame: Every 2 cycles up to 12 months until progressive disease (PD); Participants who discontinue study drug before PD: Follow-Up (FU)-every 12 weeks up to 12 months until PD/other cancer therapy; CA 125 Day 1 of cycle, End of Treatment and FU (Up to 22 Months)
Population: Response-evaluable population is defined as all participants who have measurable neoplastic disease according to the RECIST criteria OR participants with a CA 125 level > 40 units/milliliter (mL) and clinical evidence of neoplastic disease and received at least 1 dose of alisertib and have at least 1 post-baseline response assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Alisertib 50 mg (Platinum-Refractory) | Alisertib 50 mg (Platinum-Resistant)
Number analyzed (Participants) | 6 | 25
percentage of participants | 0 | 12

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time in days from the date of first study drug administration to the date of first documented Progressive Disease (PD) or death. PD is defined as 20% increase in the sum of the longest diameter of target lesions. CA 125 progression for participants with normal CA 125 levels is defined as a CA 125 level > 2 times the upper limit of normal and for participants with elevated values during the trial, is defined as a CA 125 level greater than 2 times the nadir value of CA 125. For a participant who has not progressed and has not died, PFS is censored at the last response assessment that is stable disease (SD) or better.
Time Frame: Every 2 cycles up to 12 months until PD; Participants who discontinue study drug before PD: FU - every 12 weeks up to 12 months until PD/other cancer therapy; CA 125 Day 1 of cycle, End of Treatment and FU (Up to 22 Months)
Population: Response-evaluable population is defined as all participants who have measurable neoplastic disease according to RECIST criteria OR participants with CA 125 level > 40 units/mL and clinical evidence of neoplastic disease and received at least 1 dose of alisertib and have at least 1 post-baseline response assessment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alisertib 50 mg (Platinum-Refractory) | Alisertib 50 mg (Platinum-Resistant)
Number analyzed (Participants) | 6 | 25
days | 36.5 [23.0 to 120.0] | 77.0 [43.0 to 122.0]

3. Secondary Outcome: Duration Of Response (DOR)
Description: DOR is defined as the time from the date of first documentation of a confirmed response to the date of first documented PD. PD is defined as 20% increase in the sum of the longest diameter of target lesions.
Time Frame: as for outcome 2
Population: Due to study termination, there was insufficient data to perform this analysis.
Arm/Group | Alisertib 50 mg (Platinum-Refractory) | Alisertib 50 mg (Platinum-Resistant)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time To Progression (TTP)
Description: TTP is defined as the time in days from the date of first study drug administration to the date of first documentation of PD. PD is defined as 20% increase in the sum of the longest diameter of target lesions.
Time Frame: as for outcome 2
Population: Due to study termination, there was insufficient data to perform this analysis.
Arm/Group | Alisertib 50 mg (Platinum-Refractory) | Alisertib 50 mg (Platinum-Resistant)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate is defined as the percentage of participants with response and stable disease (SD), where in order for SD to qualify as having clinical benefit, there must be no progression of neoplastic disease for at least 4 treatment cycles.
Time Frame: as for outcome 2
Population: Response-evaluable population is defined as all participants who have measurable neoplastic disease according to the RECIST criteria OR participants with a CA 125 level > 40 units/mL and clinical evidence of neoplastic disease and receive at least 1 dose of alisertib and have at least 1 post-baseline response assessment
Measure: Number; unit: percentage of participants
Arm/Group | Alisertib 50 mg (Platinum-Refractory) | Alisertib 50 mg (Platinum-Resistant)
Number analyzed (Participants) | 6 | 25
percentage of participants | 0 | 32

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events and Serious Adverse Events
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A Serious Adverse Event (SAE) A serious is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: First dose to 30 days past last dose (Up to 18.9 Months)
Population: Safety Population is defined as all participants who received any amount of alisertib.
Measure: Number; unit: participants
Arm/Group | Alisertib 50 mg (Platinum-Refractory) | Alisertib 50 mg (Platinum-Resistant)
Number analyzed (Participants) | 6 | 25
participants
  AE | 6 | 24
  SAE | 4 | 7

7. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as Treatment-Emergent Adverse Events
Description: Vital signs included blood pressure, pulse rate, and oral temperature collected throughout the study. . A treatment-emergent adverse event is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Baseline, Cycle 1 Days 8 and 15, then Day 1 of every cycle (21 days), End of Treatment, End of Study/FU every 12 weeks for up to 12 months (Up to 22 Months)
Population: Safety Population is defined as all participants who received any amount of alisertib.
Measure: Number; unit: participants
Arm/Group | Alisertib 50 mg (Platinum-Refractory) | Alisertib 50 mg (Platinum-Resistant)
Number analyzed (Participants) | 6 | 25
participants
  Pyrexia | 2 | 6
  Dyspnoea | 0 | 4
  Weight decreased | 0 | 3
  Tachycardia | 0 | 2
  Hypertension | 0 | 2
  Dyspnoea exertional | 0 | 1
  Bradycardia | 0 | 1
  Shock | 1 | 0

8. Secondary Outcome: Number of Participants With Abnormal Laboratory Values Reported as Treatment-Emergent Adverse Events
Description: Laboratory tests included Hematology and Chemistry. Abnormal laboratory value were assessed as an AE if the value leads to discontinuation or delay in treatment, dose modification, therapeutic intervention, or is considered by the investigator to be a clinically significant change from baseline. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Baseline, Cycle 1 Days 8 and 15, then Every cycle Days 1, 8 and 15 to End of Treatment Up to 18.0 Months
Population: Safety Population is defined as all participants who received any amount of alisertib.
Measure: Number; unit: participants
Arm/Group | Alisertib 50 mg (Platinum-Refractory) | Alisertib 50 mg (Platinum-Resistant)
Number analyzed (Participants) | 6 | 25
participants
  Neutropenia | 3 | 17
  Anaemia | 2 | 14
  Leukopenia | 1 | 11
  Thrombocytopenia | 1 | 8
  Dehydration | 1 | 7
  Hypokalaemia | 2 | 4
  Alanine aminotransferase increased | 0 | 6
  Aspartate aminotransferase increased | 0 | 6
  Hyperglycaemia | 1 | 4
  Hypomagnesaemia | 1 | 4
  Blood alkaline phosphatase increased | 1 | 4
  Febrile neutropenia | 0 | 3
  Hyponatraemia | 1 | 2
  Haemoglobin decreased | 1 | 2
  Granulocytopenia | 0 | 2
  Neutrophil count increased | 0 | 2
  White blood cell count increased | 0 | 2
  Hyperbilirubinaemia | 1 | 1
  Lymphopenia | 1 | 0
  Hyperkalaemia | 0 | 1
  Hypernatraemia | 0 | 1
  Hypercholesterolaemia | 0 | 1
  Transaminases increased | 1 | 0
  Granulocyte count decreased | 0 | 1
  Blood calcium increased | 0 | 1
  Blood magnesium decreased | 0 | 1
  Platelet count decreased | 1 | 0
  Blood albumin decreased | 0 | 1
  Creatinine renal clearance decreased | 0 | 1
  Hypoxia | 0 | 1
  Bacteraemia | 1 | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug to 30 past last dose of study drug (Up to18.9 Months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Alisertib 50 mg (Platinum-Refractory): Alisertib 50 mg, capsules, orally, twice daily for 7 days, followed by 14-day washout period in 21-day cycles until disease progression or unacceptable treatment-related toxicity (Up to 26 Cycles).Platinum-refractory disease is characterized by a lack of response, progression, or recurrence of disease during a course of platinum-based therapy.
Arm/Group | Alisertib 50 mg (Platinum-Refractory) | Alisertib 50 mg (Platinum-Resistant)
Serious Adverse Events (participants affected / at risk) | 4/6 | 7/25
Other Adverse Events (participants affected / at risk) | 6/6 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alisertib 50 mg (Platinum-Refractory) (N=6) | Alisertib 50 mg (Platinum-Resistant) (N=25)
Stomatitis (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal mass (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 2
Clostridium colitis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Shock (Vascular disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alisertib 50 mg (Platinum-Refractory) (N=6) | Alisertib 50 mg (Platinum-Resistant) (N=25)
Diarrhoea (Gastrointestinal disorders) | 3 | 14
Stomatitis (Gastrointestinal disorders) | 2 | 13
Nausea (Gastrointestinal disorders) | 3 | 11
Vomiting (Gastrointestinal disorders) | 4 | 8
Abdominal pain (Gastrointestinal disorders) | 2 | 8
Constipation (Gastrointestinal disorders) | 1 | 4
Ascites (Gastrointestinal disorders) | 1 | 2
Flatulence (Gastrointestinal disorders) | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 2
Abdominal rigidity (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 16
Anaemia (Blood and lymphatic system disorders) | 1 | 13
Leukopenia (Blood and lymphatic system disorders) | 1 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 7
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Fatigue (General disorders) | 3 | 15
Pyrexia (General disorders) | 1 | 5
Asthenia (General disorders) | 0 | 3
Chills (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 0 | 3
Early satiety (General disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 14
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 4
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 7
Dehydration (Metabolism and nutrition disorders) | 1 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Headache (Nervous system disorders) | 1 | 5
Somnolence (Nervous system disorders) | 0 | 4
Dizziness (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 2
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 6
Aspartate aminotransferase increased (Investigations) | 0 | 6
Blood alkaline phosphatase increased (Investigations) | 1 | 4
Haemoglobin decreased (Investigations) | 1 | 2
Weight decreased (Investigations) | 0 | 3
Neutrophil count increased (Investigations) | 0 | 2
White blood cell count increased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 3
Sinusitis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Depression (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 2
Vision blurred (Eye disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Bladder spasm (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.